CLINICAL TRIAL: NCT03751566
Title: Acupuncture as the Therapeutic Modalities of Acute Toxicity in the Radiotherapy of Head and Neck Tumors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Masaryk Memorial Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MOU-001
Record Dates: First submitted 2018-11-15; First posted 2018-11-23 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Malignant Tumor of Soft Tissue of Head, Face and Neck
MeSH Terms: conditions — Facies | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Regimen A (Active Comparator): Regimen A (control regimen): standard support treatment of adverse events of the radiotherapy.
  Interventions: Drug: Standard supportive therapy
- Regimen B (Experimental): Regimen B (acupuncture regimen): standard support treatment of adverse events of the radiotherapy and acupuncture.
  Interventions: Other: Acupuncture; Drug: Standard supportive therapy

INTERVENTIONS:
Other: Acupuncture — Schedule of the acupuncture:
  Acupuncture may be done ambulant or during hospitalisation . Acupuncture will be administered 1-3 times a week ( in case of severe toxicity and problems caused by the radiotherapy, it may continue also after the termination of the radiotherapy.) Acupuncture needles will be left for 5- 30 minutes, as per individual need of the patients.
  Acupuncture will be performed by a physician trained in acupuncture.
  Arms: Regimen B
Drug: Standard supportive therapy — Standard supportive therapy

SUMMARY:
The aim of the study is to evaluate the benefit of the acupuncture as healing modalities in the therapy of acute toxicity of radiotherapy.

DETAILED DESCRIPTION:
The study will enroll 100 patients in current radiotherapy of the head and neck cancer with acute radiotoxic symptoms at least of G1. The patients will be randomized (by ticket) in two regimens 1:1.

Regimen A (control regimen): standard support treatment of adverse events of the radiotherapy.

Regimen B (acupuncture regimen): standard support treatment of adverse events of the radiotherapy and acupuncture.

Due to the disease and patients differences, treatment will be individualized. Used acupuncture points will be documented. The patients difficulties will be observed and their medication and will be recorded in the patient diary.

Possible skin toxicities wil be documented by the photography.

Before the randomization, all subjects will sign the voluntary informed consent. After the achievement of 50 enrolled subjects in any regimen, the enrollment will continue only to the other regimen.

Head and neck cancer therapy will include only curative and adjuvant radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Curative and adjuvant radiotherapy for head and neck tumors;
* PS 1-2;
* Patient collaboration in evaluation of the toxicity diary.

Exclusion Criteria:

* Palliative radiotherapy in the head and neck tumor;
* PS 3;
* Non-compliance of the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-10-05 (Actual); Primary Completion 2023-09-04 (Actual); Study Completion 2026-10-04 (Estimated)

PRIMARY OUTCOMES:
Management of acute toxicity of radiotherapy with acupuncture: Reducing the grade of acute toxicity in radiotherapy | six months after the end of radiotherapy
  Reducing the grade of acute toxicity in radiotherapy.

SECONDARY OUTCOMES:
Management of chronic toxicity of radiotherapy with acupuncture: Lower incidence of chronic toxicity of radiotherapy | six months after the end of radiotherapy
  Lower incidence of chronic toxicity of radiotherapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Masaryk Memorial Cancer Institute, Brno, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Meng Z, Garcia MK, Hu C, Chiang J, Chambers M, Rosenthal DI, Peng H, Zhang Y, Zhao Q, Zhao G, Liu L, Spelman A, Palmer JL, Wei Q, Cohen L. Randomized controlled trial of acupuncture for prevention of radiation-induced xerostomia among patients with nasopharyngeal carcinoma. Cancer. 2012 Jul 1;118(13):3337-44. doi: 10.1002/cncr.26550. Epub 2011 Nov 9. PMID 22072272
- [Background] Braga FP, Lemos Junior CA, Alves FA, Migliari DA. Acupuncture for the prevention of radiation-induced xerostomia in patients with head and neck cancer. Braz Oral Res. 2011 Mar-Apr;25(2):180-5. doi: 10.1590/s1806-83242011000200014. PMID 21537645
- [Derived] Dymackova R, Kazda T, Slavik M, Selingerova I, Slampa P, Slama O. Acupuncture in the treatment of acute toxicity during and after head and neck cancer radiotherapy: Interim analysis of randomized prospective open-label trial. Biomed Pap Med Fac Univ Palacky Olomouc Czech Repub. 2020 Dec;164(4):454-460. doi: 10.5507/bp.2020.021. Epub 2020 Jun 18. PMID 32597419